CLINICAL TRIAL: NCT01659398
Title: Enhanced External Counterpulsation and Its Effects on Vascular Hemodynamics in Cognitively Impaired Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Patrick Moriarty, MD, FACP, FACC (Other)
Responsible Party: Sponsor-Investigator, Patrick Moriarty, MD, FACP, FACC, Director, Clinical Pharmacology, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13106
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Alzheimer's Disease; cerebral blood flow; ophthalmic blood flow; blood viscosity
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Counterpulsation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced external counterpulsation (EECP) (Experimental)
  Interventions: Device: External Counterpulsation (EECP)
- Subjects not receiving EECP (No Intervention): Control group to measure data from experimental group against.

INTERVENTIONS:
Device: External Counterpulsation (EECP) — A noninvasive neuroimaging technique. Administration of 35 hours EECP therapy over a 7 week period. EECP to be administered for 1 hour, 5 times a week.
  Arms: Enhanced external counterpulsation (EECP)

SUMMARY:
The aim of this study is to investigate whether enhanced external counterpulsation (EECP) therapy for 7 consecutive weeks will improve cerebral blood flow and possibly over time enhance or slow down breakdown of cognitive function in patients diagnosed with mild cognitive impairment (MCI).

ELIGIBILITY:
Inclusion Criteria:

* An adult between 18 and 85 years of age.
* Has been evaluated to have a CDR (Clinical Dementia Rating) Score of 0.5
* Male or female (if female must be postmenopausal for at least 1 year, surgically sterile or using an effective form of contraception).
* Able to speak and read English.
* Willing to comply with study specific instructions, and complete all study procedures according to protocol.
* Able to understand study rationale and sign informed consent.

Exclusion Criteria:

* Diagnosed with glaucoma
* History of developing adverse effects to ophthalmic dilating agents (phenylephrine or tropicamide).
* Currently taking warfarin and dabigatran (Pradaxa).
* History of having arrhythmias - can interfere with EECP triggering.
* Subject has bleeding diathesis.
* Subject has active thrombophlebitis.
* Subject has severe lower extremity vaso-occlusive disease.
* Subject has a documented aortic aneurysm requiring surgical repair.
* Subject is pregnant.
* Subject with blood pressure higher than 180/110 mmHg.
* Subject with a heart rate more than 120 bpm.
* Subject with high risk of complications from increased venous return.
* Subject with clinically significant valvular disease.
* Subjects with severe vascular disease as established by the Hachinski Ischemic Index.
* Subjects with pacemakers and other metallic implantable devices.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function | Baseline, Week 7, 6 Month
  Change in cognitive function measured using the Alzheimer's Disease Assessment Scale-cognitive sub-scale (ADAS-cog). Scale is used to determine patient's mental status. The scale has 11 parts and scores range from 0 (no impairment) to 70 (severe impairment).

SECONDARY OUTCOMES:
Change in Ophthalmic blood flow (OBF) | Baseline to Week 7
Change in Blood Viscosity | Baseline to Week 7
Cholesterol composition of the blood | Baseline to week 7

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Moriarty, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States